CLINICAL TRIAL: NCT02000466
Title: FluLaval® Quadrivalent Pregnancy Registry: a Prospective, Exploratory, Cohort Study to Detect and Describe Any Abnormal Pregnancy Outcomes in Women Intentionally or Unintentionally Vaccinated With FluLaval® Quadrivalent During Pregnancy or Within 28 Days Preceding Conception
Brief Title: FluLaval® Quadrivalent Pregnancy Registry
Status: Withdrawn | Type: Observational
Why Stopped: GSK has merged all individual pregnancy registries, which are terminated, for its seasonal influenza vaccines into one combined registry, EPI-FLU-039 VS US PR.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201086
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Influenza
Keywords: Women; Pregnancy exposure; FluLaval Quadrivalent; Pregnancy outcome; Pregnancy Registry
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Exposed cohort
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Initial and follow-up data will be collected using questionnaires

SUMMARY:
The purpose of this pregnancy registry study is to detect and describe any abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with FluLaval Quadrivalent. The Registry requires voluntary, prospective reporting of eligible pregnancies by patients and health care providers (HCPs). Data such as vaccination with FluLaval Quadrivalent during pregnancy or within 28 days preceding conception, potential confounding factors (such as exposure to other medications) and information related to the outcome of the pregnancy will be collected prospectively.

DETAILED DESCRIPTION:
Some pregnancy exposures may be reported after pregnancy outcome has been identified (retrospective reports). The Registry will capture retrospective reports, but these reports will not be included in the analyses of prospective reports.

Pregnancy outcome data will be collected using questionnaires within 3 months of the estimated date of delivery (EDD) and approximately 6 months and 12 months after the EDD from 30 November 2013 to 31 May 2018.

ELIGIBILITY:
Inclusion Criteria:

A subject will be included in the Registry if all of the following criteria are met:

* Exposure to vaccine occurs during pregnancy or within 28 days preceding conception.
* Subject is a US resident.
* A HCP is identified (name, address and phone number).
* Subject can be identified (by GSK or HCP).

Data from registered subjects will be included in the analyses if the following criterion is met:

• Pregnancy is ongoing and the outcome is unknown.

Exclusion Criteria:

Data from registered subjects will not be included in the analyses if the following criterion is met:

• Outcome of pregnancy is known at the time of initial report. Types of known outcomes include prenatal testing reports in which the results are abnormal or outside the reference range, indicating possible abnormality in the fetus. Pregnancies in which prenatal testing indicates a normal pregnancy would also be excluded because inclusion of such pregnancies could potentially bias results toward a lower overall estimate of risk for defects. Typically pregnancies > 16 weeks gestation will have undergone prenatal testing that can identify whether a child has congenital abnormalities.

Ages: 12 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women, residing in the US, exposed to FluLaval Quadrivalent and who are volunteering to take part in the Pregnancy Registry before the outcome of the pregnancy is known.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any abnormal pregnancy outcomes in women intentionally or unintentionally vaccinated with FluLaval Quadrivalent during pregnancy or within 28 days preceding conception | Up to 12 months after EDD

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline